CLINICAL TRIAL: NCT01464905
Title: A Phase 3, Multicenter, Double-blind,Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of NU100 in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: Phase 3 Study to Evaluate Efficacy and Safety of NU100 in Patients With Relapsing Remitting Multiple Sclerosis (RRMS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nuron Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-NU100-01.00
Record Dates: First submitted 2011-10-31; First posted 2011-11-04 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NU100 (Experimental)
  Interventions: Biological: NU100
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- recombinant human interferon beta- 1b (Active Comparator)
  Interventions: Biological: rhIFN beta-1b

INTERVENTIONS:
Biological: NU100 — 0.25 mg SQ, every other day for 12 months
  Arms: NU100
Biological: Placebo — 1 mL SQ, every other day for 4 months
  Arms: Placebo
Biological: rhIFN beta-1b — 0.25 mg SQ, every other day for 12 months
  Arms: recombinant human interferon beta- 1b

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of NU100 in patients with relapsing remitting multiple sclerosis (RRMS) as compared to placebo and an active comparator. The primary clinical objective selected for this Phase 3 study, the cumulative number of new combined unique active lesions (CALs; defined as new gadolinium T1-weighted lesions and non-enhancing new and newly enlarging T2-weighted lesions) on magnetic resonance imaging (MRI) scans over the course of 4 and 12 months of treatment to demonstrate the superiority of NU100 to placebo and the non-inferiority of NU100 to Betaferon®, respectively.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to participate in the study if all of the following criteria are met at both screening (V-1) and baseline (V0):

1. Female or male patients, aged between 18 and 60 years, inclusive
2. Signed and dated statement of informed consent
3. Diagnosis of RRMS according to McDonald's Criteria - revision 2010 (Polman et al., 2011)
4. Interferon (IFN) beta-1b naïve
5. Expanded Disability Status Scale (EDSS) score of < 5.5
6. At least 1 documented relapse in the past year (defined as the appearance of a new clinical sign/symptom [one that had been stable for at least 30 days] that persisted for a minimum of 24 hours in the absence of fever) ---or--- a subclinical sign/symptom (defined as a Gd-enhancing lesion or a new T2 lesion demonstrated on MRI examination on a prior MRI that has been completed within 1 year of the screening MRI). The Screening (V-1) MRI should not be used for this determination.
7. No relapse in the 4 weeks prior to the screening visit (V-1).
8. Must be in a clinically stable or improving neurological state 4 weeks preceding the screening visit (V-1).

Exclusion Criteria:

Patients meeting any of the following exclusion criteria at screening (V-1) and baseline (V0) will not be enrolled in the study:

1. Relapse at the baseline visit (V0) or occurring within 4 weeks prior to the screening visit (V-1)
2. Intake of glatiramer acetate within 3 months prior to the screening (V-1) visit
3. Intake of previous immunotherapy or immunosuppressant treatment, within 4 months prior to the screening (V-1) visit
4. Intake of or previously received therapy with cladribine or alemtuzumab
5. An active viral, bacterial, or systemic fungal infection within 1 week of baseline (V0)
6. Use of systemic steroids within 3 weeks prior to the screening (V-1) MRI
7. Progressive disease
8. Level of liver enzymes 2.5 x the upper limit of normal
9. Abnormal renal function (estimated Glomerular Filtration Rate [eGFR] < 60 ml/min/1.73 m2 )
10. Positive serology or history for Hepatitis B, C, or human immunodeficiency virus (HIV)
11. Serious or acute coronary diseases, defined by at least 1 of the following conditions:

    * Clinical symptoms of ischemic heart disease
    * ST elevation or depression > 2 mm on the electrocardiogram (ECG)
    * Clinical symptoms of cardiac failure and/or current medical treatment for cardiac failure
    * Severe ventricular arrhythmia (frequent premature ventricular beats)
    * Atrioventricular block at third level
12. Chronic use of non-steroidal anti-inflammatory drugs
13. History of any of the following:

    * Severe depression or suicide attempt
    * Uncontrolled seizure disorder
    * Cancer, excluding adequately treated basal cell carcinoma of the skin or adequately treated in situ carcinoma of the cervix
    * Previous contrast reaction to gadolinium or any other contraindications to MRI (e.g., metal in the eye, pacemakers, aneurysm clip)
14. Allergy to human albumin or to mannitol
15. Excessive alcohol use or illicit drug use
16. Women who are breast feeding, pregnant, or planning to become pregnant, or are unwilling to use an effective birth control method while on study
17. Medical, psychiatric, or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study
18. Participation in any other study involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study Current participation in other clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
New CALs after 4 months of treatment based on the MRI outcomes obtained at 4 and 12 months | 2 to 12 months
  The primary clinical objective selected for this Phase 3 study, the cumulative number of new combined unique active lesions (CALs; defined as new gadolinium T1-weighted lesions and non-enhancing new and newly enlarging T2-weighted lesions) on magnetic resonance imaging (MRI) scans over the course of 4 and 12 months of treatment to demonstrate the superiority of NU100 to placebo and the non-inferiority of NU100 to Betaferon®, respectively. Negative binomial regression will be used to compare the cumulative number of new CALs at the end of Month 4 and at the end of Month 12.

SECONDARY OUTCOMES:
Incidence of annualized relapse rates | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Goeken, M.D., Study Director — Nuron Biotech
Locations (12):
- Minsk, Belarus
- Sofia, Bulgaria
- Zagreb, Croatia
- Tbilisi, Georgia
- Budapest, Hungary
- Rome, Italy
- Beirut, Lebanon
- Warsaw, Poland
- Moscow, Russia
- Belgrade, Serbia
- Barcelona, Spain
- Kiev, Ukraine